CLINICAL TRIAL: NCT00959257
Title: The Effect of Long Term Inhaled Corticosteroids on the Risk of Cardiovascular Morbidities in Adults With Asthma :a Population Based Matched Controlled Study
Brief Title: The Effect of Long Term Inhaled Corticosteroids on the Risk of Cardiovascular Morbidities
Status: Completed | Type: Observational
Sponsor: The University of Hong Kong (Other)
Responsible Party: Dr. Wang Kwan Ling Julie, Medical Officer, Hospital Authority
Other Study IDs: UW 08-407
Record Dates: First submitted 2009-08-09; First posted 2009-08-14 (Estimated); Last update posted 2009-08-14 (Estimated); Status verified 2009-08

CONDITIONS: Asthma
Keywords: Asthma; Inhaled corticosteroids; Cardiovascular morbidities; Systemic inflammation
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Whole blood, plasma, serum and DNA
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Asthma: Asthma patients on inhaled corticosteroids
- Control: Select matched controls from the general population database of Cardiovascular Risk Factor Prevalence Study 2 (CRISPS2)

SUMMARY:
Cardiovascular disease is a major cause of morbidity and mortality worldwide. It is the second leading cause of death in Hong Kong. The disease burden is huge and effective control measures should target at prevention level. As the disease pathophysiology is linked to chronic low grade systemic inflammation, any therapeutics having the potential to reduce systemic inflammation should be vigorously explored.

The use of long-term inhaled corticosteroid (ICS) treatment in recent 2 decades has become the cornerstone in the treatment of most patients with persistent asthma with reduction in its mortality and hospital utilization. The long term safety of ICS in adults is generally very high.

Recent epidemiological studies utilizing large numbers of patients with asthma have shown that long term use of ICS is independently associated with a protective effect towards the development of myocardial infarction and cardiovascular mortality, with protective risk at 0.35 (95%CI 0.13-0.93). This effect is possibly mediated through the reduction of low grade systemic inflammation as reflected by plasma hs-CRP, from systemic absorption of the ICS.

The purpose of this study is to explore the potential protective effect of ICS on cardiovascular morbidities and its underlying link with systemic inflammation in Chinese adults with asthma compared with matched controls from the general population.

DETAILED DESCRIPTION:
Globally, cardiovascular disease is a major cause of mortality and morbidity. In the past 2 decades in Hong Kong, it has been the second leading cause of death, with death rate reaching 50/100,000 population in 2006, and the third leading cause of hospitalizations in Hospital Authority Hospitals between 2001-2005. The disease burden is huge and effective control measures should target at prevention level.

There has been substantial evidence from landmark epidemiological studies in the past 10 years that chronic low grade systemic inflammation, predominantly based on plasma hs-CRP, is an independent predictor for the development of hypertension, myocardial infarction, stroke, cardiovascular death and peripheral vascular disease. A dose-dependent risk association between hs-CRP and these cardiovascular morbidities has also been consistently demonstrated.

Asthma is a chronic inflammatory airway disorder associated with airflow obstruction and bronchial hyper-responsiveness, which affects about 10% of population in Hong Kong. It is a major respiratory disease in Hong Kong that carries significant morbidity and high hospitalization burden in all ages. The use of long-term inhaled corticosteroid (ICS) treatment in recent decades has become the cornerstone in the treatment of most patients with persistent asthma with reduction in its mortality and hospital utilization. The ultimate goal of treatment is to achieve optimal control of airway inflammation and to reduce mortality and morbidity.

Although the pathogenesis of asthma is incompletely understood, studies have shown that it is associated airway inflammation and a state of increased free radical formation, because cells derived from airways and peripheral blood of patients with asthma generate increased amount of reactive oxygen species, the level of which is related to severity of asthma. Recent preliminary studies have indicated that, apart from the presence of chronic airway inflammation, asthma may also be associated with chronic low grade systemic inflammation and increased oxidative stress. Intuitively, this asthma-related systemic inflammation may increase the risk for development of cardiovascular and cerebrovascular diseases.

Despite the propensity of asthma towards cardiovascular morbidity, recently, several epidemiological studies utilizing large numbers of patients with asthma have shown that long term use of ICS is independently associated with a protective effect towards the development of myocardial infarction and cardiovascular mortality, with protective risk at 0.35 (95%CI 0.13-0.93). This effect is possibly mediated through the reduction of low grade systemic inflammation as reflected by plasma hs-CRP from systemic absorption of the ICS.

This potential effect of ICS on reduction of chronic low grade systemic inflammation has an invaluable implication for its future application as a preventive medicine against the development of cardiovascular morbidities and mortality, especially in high risk patients.

ICS have been launched for more than 20 years, and is currently the first-line treatment for asthma. Their systemic side effects are much less than that of oral corticosteroids. Long term safety of ICS in adults is generally very high, but mild increases in risk of osteoporosis, cataracts and glaucoma have been reported in patients with high dose ICS use.

The purpose of this study is to explore the potential protective effect of ICS on cardiovascular morbidities and its underlying link with systemic inflammation in Chinese adults with asthma compared with matched controls from the general population.

ELIGIBILITY:
Inclusion Criteria:

* Adult Chinese asthma patients
* Stable persistent asthma who are current inhaled corticosteroid users OR
* Healthy controls will be non inhaled corticosteroid users matched for age, gender and BMI from the Hong Kong Cardiovascular Risk Factor Prevalence Study II (CRISPSII) carried out on a random population sample in Hong Kong

Exclusion Criteria:

* On maintenance oral steroid
* Systemic steroid use in recent 6 months
* Asthma exacerbation (GINA criteria) in recent 1 month (ie daytime or nocturnal symptoms increment, detectable wheezing on physical examination, drop in peak flow rate, drop in spirometry indexes, increase in asthma medication, emergency medical attendance for asthma, days off work for asthma etc)
* Inhaled corticosteroid use for < 6 months
* Pregnancy

Ages: 35 Years to 74 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Asthma patients will be recruited from asthma clinics of 4 centres in Hong Kong, including Queen Mary Hospital, Queen Elizabeth Hospital, Kowloon Hospital and Kwong Wah Hospital.
  Matched controls at 1:1 ratio from the general population database of Cardiovascular Risk Factor Prevalence Study II (CRISPSII) will be selected. Matching critera: age +/-5 years; same gender and BMI+/-10%.
Sampling Method: Non-Probability Sample
Enrollment: 1394 (Actual)
Dates: Start 2009-01; Primary Completion 2009-07 (Actual); Study Completion 2009-07 (Actual)

PRIMARY OUTCOMES:
Estimated prevalence and prevalence OR of cardiovascular morbidites in asthma patients using ICS expressed in 95% confidence interval | 1 year

SECONDARY OUTCOMES:
Cumulative dose response relationship and effect modification of ICS on the OR of cardiovascular morbidities, 95% confidence interval | 1 year
Cumulative Inhaled corticosteroids dose effect on the levels of hs-CRP. Adjusted change in level of hs-CRP in relation to change in ICS dosage, expressed in median and interquartile range | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Kwan-ling Julie Wang, Principal Investigator — Hospital Authority
Locations (4):
- Hong Kong (4):
  - Kowloon Hospital, Hong Kong
  - Kwong Wah Hospital, Hong Kong
  - Queen Elizabeth Hospital, Hong Kong
  - Queen Mary Hospital, Hong Kong